CLINICAL TRIAL: NCT02848846
Title: NEurocontrolled BIdirectional Artificial Upper Limb and Hand prosthesiS
Acronym: NEBIAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paolo Maria Rossini (Other)
Responsible Party: Sponsor-Investigator, Paolo Maria Rossini, Full Professor, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FP7- ICT-2013.9.6
Record Dates: First submitted 2016-06-23; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Sensorized Hand Prosthesis
Keywords: Amputees

ARMS (1):
- Robotic Hand (Experimental): The two patient enrolled will perform the task requiring the use of the robotic hand.
  Interventions: Device: Robotic Hand

INTERVENTIONS:
Device: Robotic Hand — The patients will use the robotic hand for a period of one year that will be divided in 3 different phases. The first phase is the intensive phase where the patient will use the robotic hand from Monday to Friday all days. This phase will last 6 weeks. The second phase is the semi-intensive where the patient will use the robotic hand only two days per week. This phase will last 6 weeks. The third phase is the monitoring where the patient will use the robotic hand only one day per week until the end of the trial.
  During this phases the patient will perform different task requiring the use of the robotic hand.

SUMMARY:
The NEBIAS ("NEurocontrolled BIdirectional Artificial upper limb and hand prosthesiS") proposal aims at developing and clinically evaluating (in selected amputees) a neuro-controlled upper limb prosthesis intuitively controlled and felt by the amputee as the natural one. This will be possible by means of a novel neural interface able to provide a stable and very selective connection with the nervous system. This goal will be achieved by combining microtechnology and material science and will allow, on one side, recording of the motor-related signals governing the actions of the amputated hand/arm for the motion control of a mechanical prosthesis, and on the other providing sensory feedback from tactile and kinesthetic sensors through neuromorphic stimulation of the adequate afferent pathway within the residual limb. The NEBIAS proposal is also aimed at finding out the 'language' intrinsically linking central nervous system with peripheral nerve signals in order to govern simple and complex hand/fingers movements. To reach this goal, a variety of techniques exploring brain and nerve functions will be assembled and integrated; this includes the analysis of electromagnetic brain and nerve signals, as well as of movement-related changes in brain's blood flow/metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Adult man or woman >18 yrs and < 71 yrs.
* Transradial amputation or Congenital Hand Hypoplasia
* Amputation in the chronic stable phase
* Good functionality of muscles of the stump
* Absence of severe stump pain (VAS<3)

Exclusion Criteria:

* Cognitive impairment
* Current or prior psychological impairments: Major personality disturbance (i.e. borderline, antisocial), Major depression, Bipolar I
* Pregnancy
* History of or active substance abuse disorder
* Acquired brain injury with residual impairment
* Intellectual Disability (IQ < 70)
* Prior neurological or musculo-skeletal disease
* Current or prior dermatological conditions
* Excessive sensitivity to electrical stimulation (people afraid of electrical stimulation or pain)
* Persons with other diseases that may affect the function of the nervous system. (Diabetes, HIV, Renal Failure)
* Persons with pacemakers
* People affected by autoimmune and chronic infective diseases in treatment with immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
performance of the robotic hand | 1 year
  Different level of pressure (percentage of success);
performance of the robotic hand | 1 year
  Virtual egg test (percentage of success);
performance of the robotic hand | 1 year
  Pick and Lift (percentage of success);
performance of the robotic hand | 1 year
  Texture recognition (percentage of success);
performance of the robotic hand | 1 year
  Shape recognition (percentage of success);
performance of the robotic hand | 1 year
  Compliance recognition (percentage of success)

SECONDARY OUTCOMES:
Cortical map changes | 1 year
  Primary motor area (change of dimension and shape);
Cortical map changes | 1 year
  Primary somatosensory area (change of dimension and shape);

CONTACTS AND LOCATIONS:
Overall Officials: paolo m rossini, professor, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Fondazione Policlinico Agostino Gemelli, Rome, Lazio, Italy

REFERENCES:
- [Derived] Cracchiolo M, Panarese A, Valle G, Strauss I, Granata G, Iorio RD, Stieglitz T, Rossini PM, Mazzoni A, Micera S. Computational approaches to decode grasping force and velocity level in upper-limb amputee from intraneural peripheral signals. J Neural Eng. 2021 Apr 6;18(5). doi: 10.1088/1741-2552/abef3a. PMID 33725672
- [Derived] Valle G, D'Anna E, Strauss I, Clemente F, Granata G, Di Iorio R, Controzzi M, Stieglitz T, Rossini PM, Petrini FM, Micera S. Hand Control With Invasive Feedback Is Not Impaired by Increased Cognitive Load. Front Bioeng Biotechnol. 2020 Apr 3;8:287. doi: 10.3389/fbioe.2020.00287. eCollection 2020. PMID 32318562